CLINICAL TRIAL: NCT00826176
Title: A Multi-center, Open Label Trial, to Show Efficacy and Safety of 4.0 mg.Kg-1 Sugammadex Administered at a Depth of Neuromuscular Blockade of 1-2 PTC Induced by Rocuronium in Chinese and European ASA I-III Subjects Undergoing Elective Surgery Under Propofol Anesthesia
Brief Title: Efficacy and Safety of 4.0 mg/kg Sugammadex at 1-2 PTC in Chinese and European Subjects (Study 19.4.335)(P05775AM1)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05775; 19.4.335
Record Dates: First submitted 2009-01-15; First posted 2009-01-21 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Anesthesia, General; Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex in Caucasian Subjects (Experimental): At 1-2 post-tetanic counts (PTC) after the last dose of rocuronium, 4.0 mg.kg-1 sugammadex was to be administered. Caucasian subjects living in Europe.
  Interventions: Drug: Sugammadex
- Sugammadex in Chinese Subjects (Experimental): At 1-2 post-tetanic counts (PTC) after the last dose of rocuronium, 4.0 mg.kg-1 sugammadex was to be administered. Chinese subjects living in China.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — After induction of anesthesia an intubation dose of 0.6 mg/kg rocuronium was to be administered. Maintenance doses of 0.1-0.2 mg/kg rocuronium intravenous (IV) could have been administered if necessary. At 1-2 PTC after the last administration of rocuronium, an IV single bolus dose of 4.0 mg/kg sugammadex was to be administered.
  Other Names: Org 25969, Bridion®

SUMMARY:
The present trial is set up to evaluate the efficacy and safety of 4.0 mg.kg-1 sugammadex in Chinese and Caucasian subjects for registration purposes in China.

ELIGIBILITY:
Inclusion Criteria:

-Subjects who are willing to provide informed consent; be between 18 and 64 years old; are American Society of Anaesthesiology (ASA) class 1-3 (extremes included); scheduled for elective surgery under general anesthesia, allowing stable neuromuscular monitoring, which requires neuromuscular blockade using

rocuronium; be compliant with the dose/visit schedules, and use an accepted method of contraception (if applicable).

For China only: Subjects of Chinese descent born in China, never emigrated out of China and have a Chinese home address. For Europe only: Subjects of Caucasian descent born in Europe, never emigrated out of Europe and have a European home address.

Exclusion Criteria:

-Subjects with expected difficult intubation, neuromuscular disorders affecting neuromuscular blockade, significant renal/hepatic dysfunction, use of a tourniquet, (family) history of malignant hyperthermia, allergy to general anesthesia medications, contraindication to study drugs, breast feeding, pregnant, participation in previous or new trials, a clinically significant condition that may interfere with the trial, or membership in the

(family of) study/sponsor staff.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

REFERENCES:
- [Result] Yu B, Wang X, Helbo Hansen HS, Huang W-Q, Askeland B, Li S, Ding Z, Abels E, Rietbergen H, Woo T, Pendeville P. Sugammadex 4.0 mg/kg reversal of deep rocuronium-induced neuromuscular blockade: a multicenter study in Chinese and Caucasian patients. J Anesthe Clin Res. 2014;5:408. doi: 10.4172/2155-6148.1000408

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were screened but not enrolled (one Chinese subject and one Caucasian subject).
Period: Overall Study
Arm/Group | Sugammadex in Chinese Subjects | Sugammadex in Caucasian Subjects
Started | 128 (enrolled) | 36 (enrolled)
Completed | 115 (treated and completed) | 36 (treated and completed)
Not Completed | 13 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject Withdrew Consent | 3 | 0
Not completed — Administrative | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex in Chinese Subjects | Sugammadex in Caucasian Subjects | Total
Number analyzed (Participants) | 115 | 36 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (10.0) | 47.2 (11.0) | 47.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 29 | 95
  Male | 49 | 7 | 56

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of Sugammadex to Recovery of the T4/T1 Ratio to 0.9
Description: Neuromuscular functioning was monitored by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. Nerve stimulation continued until the ratio of the magnitude of the fourth twitch (T4) to first twitch (T1) reached at least 0.9. The greater the T4/T1 ratio the greater the recovery from neuromuscular blockade, with a value of 1.0 representing full recovery.
  Analysis of recovery in Chinese subjects was the primary objective; Caucasian subjects and between-group analyses were secondary.
Time Frame: Start of administration of sugammadex to recovery from neuromuscular blockade
Population: The Full Analysis Set (FAS) consisted of all subjects who received sugammadex and had at least one efficacy measurement. One treated Chinese subject did not have any efficacy data and was thus excluded from the FAS. Hence, 114 Chinese Asian and 36 European Caucasian subjects were included in the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex in Chinese Subjects | Sugammadex in Caucasian Subjects
Number analyzed (Participants) | 114 | 36
minutes | 2.3 [2.1 to 2.6] | 1.4 [1.3 to 1.6]
Statistical Analysis 1: Comparison: Sugammadex in Chinese Subjects; Test type: Superiority or Other; upper limit of tolerance interval (min.) = 6.4 — The tolerance interval (TI) refers to a fixed proportion (in this trial set to 95%) of the population with a stated confidence (in this trial, 95%). Efficacy was to be claimed in case the upper limit of TI was below the prespecified margin of 10 min
Statistical Analysis 2: Comparison: Sugammadex in Caucasian Subjects; Test type: Superiority or Other; upper limit of tolerance interval (min.) = 3.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Sugammadex in Chinese Subjects vs Sugammadex in Caucasian Subjects; Test type: Non-Inferiority or Equivalence — Equivalence between the two subject populations was to be claimed in the event that the two-sided 95% confidence interval was entirely within the interval ranging from -60 to +60 seconds; median difference (seconds) = 49, 95% CI [30 to 72] — The estimated median difference (Chinese minus Caucasian) in time to recovery of the T4/T1 ratio to 0.9

2. Secondary Outcome: Time From Start of Administration of Sugammadex to Recovery of the T4/T1 Ratio to 0.7
Description: Neuromuscular functioning was monitored by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. The greater the T4/T1 ratio the greater the recovery from neuromuscular blockade.
Time Frame: Start of administration of sugammadex to recovery from neuromuscular blockade
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex in Chinese Subjects | Sugammadex in Caucasian Subjects
Number analyzed (Participants) | 114 | 36
minutes | 1.6 [1.5 to 1.8] | 1.1 [1.0 to 1.2]

3. Secondary Outcome: Time From Start of Administration of Sugammadex to Recovery of the T4/T1 Ratio to 0.8
Description: as for outcome 2
Time Frame: Start of administration of sugammadex to recovery from neuromuscular blockade
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex in Chinese Subjects | Sugammadex in Caucasian Subjects
Number analyzed (Participants) | 114 | 36
minutes | 1.9 [1.7 to 2.1] | 1.2 [1.1 to 1.3]

ADVERSE EVENTS:
Arm/Group | Sugammadex in Chinese Subjects | Sugammadex in Caucasian Subjects
Serious Adverse Events (participants affected / at risk) | 0/115 | 1/36
Other Adverse Events (participants affected / at risk) | 46/115 | 20/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex in Chinese Subjects (N=115) | Sugammadex in Caucasian Subjects (N=36)
post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex in Chinese Subjects (N=115) | Sugammadex in Caucasian Subjects (N=36)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 6 (9)
abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 6 (10)
nausea (Gastrointestinal disorders) | 8 (8) | 7 (10)
vomiting (Gastrointestinal disorders) | 12 (12) | 5 (5)
instillation site erythema (General disorders) | 0 (0) | 2 (2)
incision site pain (Injury, poisoning and procedural complications) | 26 (26) | 1 (1)
procedural hypotension (Injury, poisoning and procedural complications) | 3 (3) | 6 (10)
wound complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (7)
dizziness (Nervous system disorders) | 3 (3) | 5 (8)
cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1)
rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may not publish/publicly present interim results without prior consent of Sponsor. Any materials that report results of the study must be sent to Sponsor 45 days prior to submission for publication/presentation. Sponsor has right to review and comment. In case of any disagreements concerning appropriateness of the materials, investigator and Sponsor must meet to make a good faith effort to discuss/resolve the issues or disagreement, prior to submission for publication/presentation.